CLINICAL TRIAL: NCT02233179
Title: Body-worn Sensor Technology for Improving Diabetic Care During Activities of Daily Living
Brief Title: The Association Between Unprotected Standing, Walking and Wound Healing in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Qatar National Research Foundation, Qatar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0900000701
Record Dates: First submitted 2014-08-08; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Removable Cast Walker (Experimental): An offloading device that can be removed by the patients
  Interventions: Device: Removable cast walker
- Irremovable Cast Walker (Active Comparator): A removable cast rendered irremovable using instant total contact cast, so patients cannot remove offloading device.
  Interventions: Device: Irremovable cast walker

INTERVENTIONS:
Device: Removable cast walker — Offloading device that can be removed by patients.
  Other Names: Cast walker from Ossur, Reykjavik, Iceland
  Arms: Removable Cast Walker
Device: Irremovable cast walker — Offloading device that cannot be removed by patients.
  Other Names: Cast walker from Ossur, Reykjavik, Iceland
  Arms: Irremovable Cast Walker

SUMMARY:
The aim of the study was to explore the association between activities of daily living ( measured using a body-worn sensor) on wound healing in diabetic patients. Since this was an exploratory study, there was no study hypothesis.

DETAILED DESCRIPTION:
Diabetes patients with active foot ulcers were recruited and monitored for activities of daily living while wearing an offloading device.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older with non-infected, non-ischemic foot ulcers
* active neuropathic foot ulcer

Exclusion Criteria:

* major foot amputation
* active Charcot arthropathy
* ankle brachial index of 0.5 or less
* history of substance abuse within 6 months
* inability to walk 20m

Ages: 37 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Wound size | 12 weeks
  Wound size was measured every week for 12 weeks
Daily Physical Activities | 12 weeks
  Recorded using a body-worn sensor and measured every 4 weeks for 2 days.

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- University Medical Center, Tucson, Arizona, United States